CLINICAL TRIAL: NCT02434029
Title: Double-blind, Randomized, Placebo-controlled, Phase III Trial on the Efficacy and Tolerability of a 6-week Treatment With Budesonide Effervescent Tablets vs. Placebo for Induction of Clinico-pathological Remission in Adult Patients With Active Eosinophilic Esophagitis
Brief Title: Budesonide Orodispersible Tablet vs. Placebo in Active Eosinophilic Esophagitis
Acronym: EOS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUL-1/EEA; 2014-001484-12 (EudraCT Number)
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide (Experimental): Budesonide 1mg orodispersible tablet twice daily
  Interventions: Drug: Budesonide 1mg orodispersible tablet twice daily
- Placebo (Placebo Comparator): Placebo orodispersible tablet twice daily
  Interventions: Drug: Placebo orodispersible tablet twice daily

INTERVENTIONS:
Drug: Budesonide 1mg orodispersible tablet twice daily
  Arms: Budesonide
Drug: Placebo orodispersible tablet twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to prove the superiority of a 6-weeks treatment with budesonide effervescent tablets versus placebo for the induction of clinico-pathological remission in patients with acute eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Male or female patients, 18 to 75 years of age,
* Confirmed clinico-pathological diagnosis of eosinophilic esophagitis (EoE) according to established diagnostic criteria
* Active symptomatic and histological EoE,
* A documented trial with proton pump inhibitors (PPIs) in order to rule out PPI-responsive esophageal eosinophilia,
* Negative pregnancy test in females of childbearing potential at baseline visit.

Exclusion Criteria:

* Clinical and endoscopic signs of gastroesophageal reflux disease (GERD),
* History of abnormal results in case of an optionally performed pH-monitoring of the distal esophagus,
* Patients with PPI-responsive esophageal eosinophilia
* Achalasia, scleroderma esophagus, or systemic sclerosis,
* Other clinically evident causes than EoE for esophageal eosinophilia,
* Any concomitant esophageal disease and relevant gastro-intestinal disease (celiac disease, inflammatory bowel disease, oropharyngeal or esophageal bacterial, viral, or fungal infection [candida esophagitis]),
* Any relevant systemic disease (e.g., AIDS, active tuberculosis),
* If careful medical monitoring is not ensured: cardiovascular disease, diabetes mellitus, osteoporosis, active peptic ulcer disease, glaucoma, cataract, or infection,
* Liver cirrhosis or portal hypertension,
* History of cancer in the last five years,
* History of esophageal surgery at any time or of esophageal dilation procedures within the last 8 weeks prior to screening visit,
* Upper gastrointestinal bleeding within 8 weeks prior to screening visit,
* Existing or intended pregnancy or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2016-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of clinico-pathological remission | 6 weeks

SECONDARY OUTCOMES:
Rate of patients with histological remission | 6 weeks
Rate of patients with resolutions of symptoms measured by numerical rating score of symptoms | week 6

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Mueller, PhD, Study Director — Dr. Falk Pharma GmbH
Locations (1):
- Center for Digestive Diseases Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Straumann A, Lucendo AJ, Miehlke S, Vieth M, Schlag C, Biedermann L, Vaquero CS, Ciriza de Los Rios C, Schmoecker C, Madisch A, Hruz P, Hayat J, von Arnim U, Bredenoord AJ, Schubert S, Mueller R, Greinwald R, Schoepfer A, Attwood S; International EOS-2 Study Group. Budesonide Orodispersible Tablets Maintain Remission in a Randomized, Placebo-Controlled Trial of Patients With Eosinophilic Esophagitis. Gastroenterology. 2020 Nov;159(5):1672-1685.e5. doi: 10.1053/j.gastro.2020.07.039. Epub 2020 Jul 25. PMID 32721437
- [Derived] Lucendo AJ, Miehlke S, Schlag C, Vieth M, von Arnim U, Molina-Infante J, Hartmann D, Bredenoord AJ, Ciriza de Los Rios C, Schubert S, Bruckner S, Madisch A, Hayat J, Tack J, Attwood S, Mueller R, Greinwald R, Schoepfer A, Straumann A; International EOS-1 Study Group. Efficacy of Budesonide Orodispersible Tablets as Induction Therapy for Eosinophilic Esophagitis in a Randomized Placebo-Controlled Trial. Gastroenterology. 2019 Jul;157(1):74-86.e15. doi: 10.1053/j.gastro.2019.03.025. Epub 2019 Mar 26. PMID 30922997